CLINICAL TRIAL: NCT01259518
Title: A Phase I Dose Escalation Study on the Tolerability and Activity of TriN 2755 in Patients With Advanced Solid Tumors and Sarcomas Using Two Different Dosage Regimens
Brief Title: Dose Escalation Study of TriN2755 in Advanced Solid Tumors and Sarcomas
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Trin Therapeutics GmbH (Industry)
Collaborators: University Hospital, Essen (Other); Central European Society for Anticancer Drug Research (Other); Assign Data Management and Biostatistics GmbH (Other)
Responsible Party: Georg Ludwig Managing Director, Trin Therapeutics GmbH
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIN2755-I-01
Record Dates: First submitted 2010-11-24; First posted 2010-12-14 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Once monthly administration of TRIN2755 (Experimental)
  Interventions: Drug: TRIN2755
- Once weekly administration of TRIN2755 (Experimental)
  Interventions: Drug: TRIN2755

INTERVENTIONS:
Drug: TRIN2755 — In treatment schedule A (Group A), the planned starting dose to be investigated is 25 mg TriN 2755 given once followed by a recovery period of 4 weeks. Subsequent patients can only be included on a new dose level when the safety review from all patients included at the preceding dose level(s) at Day 28 after infusion (end of Cycle 1) does not indicate relevant toxicity.
  Arms: Once monthly administration of TRIN2755
Drug: TRIN2755 — In treatment schedule B (Group B), the starting dose to be investigated is 800mg, given once every 7 days in a 4 week cycle. Subsequent patients can only be included on a new dose level when the safety review from all patients included at the preceding dose level(s) at Day 28 after the start of the first infusion (end of Cycle 1) does not indicate relevant toxicity.
  Arms: Once weekly administration of TRIN2755

SUMMARY:
This is an open-label, parallel-group, two-center, safety, activity and pharmacokinetic study of TriN 2755 given at increasing dose levels as intravenous infusions administered over 4 hours. The study is divided into two parts: Part I a dose escalation phase and Part II an extension phase.

DETAILED DESCRIPTION:
Classical chemotherapeutic agents include the class of alkylating agents with covalent modification of biopolymers and in particular, bases of DNA, as proposed mechanism of cytotoxic action. Bifunctional alkylating agents, which yield inter- or intrastrand cross-links include nitrogen mustards, mitomycin C and platinum complexes. In contrast, monofunctional alkylating agents act by reacting with single electron-rich sites in bases of DNA strands. The most prominent class of the latter group is the triazene, which is based on nitrogen-rich chemistry. It is generally accepted that triazenes, upon metabolic activation via N demethylation, yield highly reactive carbocations, which covalently bind to biopolymers. The novel triazene TriN 2755 differs from other triazenes through its physicochemical properties such as high hydrophilicity and photostability, and in particular by its potent, dose dependent antitumor activity in a spectrum of cancers including dacarbazine-resistant tumors, where treatment options for metastatic disease are still not satisfactory and medical needs exist.

This is an open-label, parallel-group, two-center, safety, activity and pharmacokinetic study of TriN 2755 given at increasing dose levels as intravenous infusions administered over 4 hours. The study is divided into two parts: Part I a dose escalation phase and Part II an extension phase.

Part I of the Study (Dose Escalation Phase):

In the first part of the study, two treatment schedules will be investigated in parallel:

Treatment schedule A: The study medication will be infused once every 28 days in a 4-week cycle (Group A) Treatment schedule B: The study medication will be infused once every 7 days in a 4-week cycle (Group B)

In treatment schedule A (Group A), the planned starting dose to be investigated is 25 mg TriN 2755 given once followed by a recovery period of 4 weeks. Subsequent patients can only be included on a new dose level when the safety review from all patients included at the preceding dose level(s) at Day 28 after infusion (end of Cycle 1) does not indicate relevant toxicity.

In treatment schedule B (Group B), the planned starting dose to be investigated is 800mg, given once every 7 days in a 4 week cycle. Subsequent patients can only be included on a new dose level when the safety review from all patients included at the preceding dose level(s) at Day 28 after the start of the first infusion (end of Cycle 1) does not indicate relevant toxicity.

Plasma samples to evaluate the pharmacokinetics of TriN 2755 are collected at predefined schedules after the first administration at each dose level and at pre-dose and at expected peak times during the subsequent administrations within the first treatment cycle only (Group B). Urine samples are collected over 24 hours after the first administration at each dose level within the first treatment cycle only.

Once the MTD is reached, two expanded cohorts of patients are treated with the Maximum Recommended Dose (MRD) which is one dose level below the MTD or at lower dose levels, if indicated. This second part of the study (expansion) allows for enrolment of approximately additional 9 patients per treatment schedule, at the chosen dose, in order to better assess the safety and possible antitumor activity of TriN 2755. The exact number of patients to be enrolled in this expanded phase is decided by a Monitoring Board. The patients are treated at or near the planned phase II dose, without expanding or prolonging the study excessively.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of age > 18 years
* Patients with a histologically / cytologically confirmed diagnosis of advanced solid tumor or sarcoma for which a treatment of proven efficacy does not exist or an established treatment(s) had failed
* Measurable or non-measurable disease according to RECIST v1.0 criteria. Patients should have at least one measurable lesion or disease which is non-measurable but can clearly be evaluated for response
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* Life expectancy of at least 3 months
* Ability to understand the nature of the study and willingness to sign a written informed consent document
* Willingness and ability to comply with the study protocol for the duration of the study

Exclusion Criteria:

* Any lymphoma or other hematological tumors
* Known brain metastases
* Earlier history of other tumors, except non melanoma-skin cancer or in situ cervical carcinoma curatively excised
* Major surgery within 4 weeks prior to treatment start
* Extensive radiotherapy, within 2 weeks of treatment start, or cytotoxic chemotherapy or limited radiotherapy within 2 weeks of treatment start
* Unresolved toxicity from prior chemotherapy (including approved and experimental drugs)
* Any of the following abnormal baseline hematological values:
* Hb < 10g/dl,
* WBC < 3.0 x 109/l Neutrophils < 1.5 x 109/l
* Platelets < 100 x 109/l
* Any of the following abnormal baseline liver function tests:
* Serum bilirubin > 1.5 x upper normal limit, > 3 x if due to tumor
* ALAT and/or ASAT > 2.5 x upper normal limit, > 5 x if due to tumor
* The following abnormal baseline renal function test:
* Serum creatinine > 1.5 mg/dl
* Creatinine clearance < 50 ml/min
* All clinically relevant cardiovascular abnormalities (i.e. myocardial infarction within the prior 6 months, cardiac arrhythmia requiring medication, uncontrolled hypertension, abnormal cardiac function (* class II of NYHA classification), cardiac failure or non compensated active heart disease (* class II of NYHA classification)
* Neurologic: symptomatic motor or sensory neurotoxicity grade 2 NCI CTC
* Primary tumor associated with central nervous system-related symptoms interfering with the informed consent or with the study
* History of psychiatric disabilities, seizures or central nervous system disorders, which is considered to be clinically significant by the investigator and could interfere with informed consent or adequate follow-up
* Major fluid effusions (e.g. ascites, pleural effusion), or clinically relevant blood loss
* Interstitial pneumonia or lung fibrosis
* History or presence of thromboses or clotting disorders
* Concomitant medication for non-vital indications with known hepatotoxic or nephrotoxic potential (e.g, aminoglycoside antibiotics)
* Serious (Grade 3-4) uncontrolled intercurrent infections
* Any history of alcohol abuse or drug addiction
* Positive results of virus serology tests (i.e. detection of HBsAg and antibodies to HCV, HIV1, HIV2, CMV and EBV)
* Clinical conditions equal to protocol definitions of DLT
* Participation in any investigational drug study within 30 days preceding treatment start
* Male or pre-menopause female patients unable to practice a medically approved method of contraception during the study and the 3-month period thereafter (all patients potentially fertile)
* Pregnancy or breast feeding women
* Any condition which in the judgment of the investigator would place the subject at undue risk or interfere with the results of the study (e.g. increased medical risks due to non malignant organ or systemic disease or secondary effects of cancer)
* History of allergic reactions attributed to compounds of the same chemical class (dacarbazine, temozolomide) as TriN 2755 or any excipients of IMP
* Mental handicap or legal incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-09 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | at baseline and beginning of every cycle

SECONDARY OUTCOMES:
Objective response rate (ORR); RECIST v1.0 Criteria | 3 Years
Progression free survival (PFS) | 3 years
Overall survival (OS) within 12 months after the first infusion of TriN 2755 | 12 months
Pharmacokinetics of TRIN2755 and its metabolites | 4 weeks
  TriN 2755 and a selection of assumed metabolites in plasma and urine samples will be analyzed by using a validated Reverse-Phase High Performance Liquid Chromatography (RV-HPLC) procedure with Mass Spectrometric (MS) detection of e.g. area únder curve(AUC) , Concentration maximum (Cmax)
Concentration of DNA methyl adducts in leucocytes and urine, analysis of DNA strand breaks | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Max E Scheulen, PHD MD, Principal Investigator — Department of Internal Medicine West German Cancer Centre University Hospital Essen Essen, Germany
Locations (1):
- Department of Internal Medicine West German Cancer Centre University Hospital Essen, Essen, Germany